CLINICAL TRIAL: NCT06616051
Title: Study Protocol for a Randomized Controlled Trial Investigating the Effectiveness of mHealth-Based Vision Screening on Uptake of Referral Services Among Children of Government Schools in Rawalpindi, Pakistan
Brief Title: Frequency of Visual Impairment Among School Children and Effectiveness of mHealth Referral Reminder on Uptake of Referral Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syed Fawad Mashhadi (Other)
Responsible Party: Sponsor-Investigator, Syed Fawad Mashhadi, Professor and Head of the department, community medicine and public health, Army medical college, Rawalpindi Medical College
Organization: Rawalpindi Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: vision320rct
Record Dates: First submitted 2024-09-22; First posted 2024-09-27 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Visual Impairment; Refractive Error
Keywords: visual impairment; mhealth; refractive error; referral reminder
MeSH Terms: conditions — Vision Disorders; Refractive Errors

STUDY DESIGN:
Intervention Model Description: This study is a Concurrent parallel group, single blinded Randomized Control Trial with 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Masking Description: The individual responsible for follow-up contacts will remain blinded to group allocation by working from a coded participant list that does not identify arm membership and will record outcomes using participant IDs only. The data analyst will receive a de-identified dataset with intervention arm masked to permit unbiased analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Parents or guardians in the intervention group will receive a multicomponent SMS reminder in addition to printed referral forms. These reminders will be delivered every Sunday, Tuesday and Thursday for a duration of eight weeks, or until the child attends the hospital. Research team has already developed an automated text message reminder system for this study, taking into account the local context. The content of the messages was designed with input from a panel of public health consultants and research supervisors, drawing on resources from the WHO Health Promotion and Disease Prevention Messages Library [21].
  Messages will be sent in Urdu, the native language, and will not require a reply. Each message will include four elements: Health promotion message, visual depiction of a child's vision, a customized action plan detailing how to get to the hospital including the location, how much money is needed and what to carry with them.
  Interventions: Other: Multicomponent SMS reminder
- Control arm (No Intervention): Among control arm, the participants screened positive for visual impairment in the control group will receive a referral form. There will be no mHealth referral reminder sent to the identified visual impaired children.

INTERVENTIONS:
Other: Multicomponent SMS reminder — SMS reminder will be delivered every Sunday, Tuesday and Thursday for a duration of eight weeks, or until the child attends the hospital. Research team has already developed an automated text message reminder system for this study, taking into account the local context. The messages was designed with input from a panel of public health consultants and research supervisors, drawing on resources from the WHO Health Promotion and Disease Prevention Messages Library [21].
  It will comprise two main components: a) web-based application for children registration and automated reminder scheduling, and b) an SMS application for text messaging that is sent automatically. Messages will be sent in Urdu, the native language, and will not require a reply. Each message will include four elements: Health promotion message, visual depiction of a child's vision, a customized action plan detailing how to get to the hospital including the location, how much money is needed and what to carry with them.
  Arms: Intervention arm

SUMMARY:
This study tested whether mobile health (mHealth) tools can affect referral uptake among schoolchildren with vision problems.Visual impairment in children often goes untreated in low- and middle-income countries, even when detected during school screenings, because parents do not follow up on referral advice.

In this randomized controlled trial, children aged 5-15 years from two government schools in Rawalpindi, Pakistan, were screened for vision problems using a smartphone-based application. Those identified with possible impairment were randomly assigned to one of two groups. The control group received the usual printed referral form, while the intervention group received the printed referral plus automated, multicomponent SMS reminders in the local language. These reminders included health promotion messages, a visual depiction of the child's vision, and practical instructions about how to reach the hospital.

The main outcome was the proportion of referred children who attended the hospital within eight weeks. Secondary analysis examined whether referral uptake was linked with child and family characteristics such as age, sex, and parental education.

This was a minimal-risk, school-based trial with 80 participants. The study was ethically approved by the Army Medical College Ethics Review Committee (NUMS). Findings are expected to provide new evidence on the usefulness of mobile phone-based reminders for improving eye health care among children in resource-limited settings.

DETAILED DESCRIPTION:
This randomized controlled trial was conducted to evaluate the effectiveness of a mobile health (mHealth)-based vision screening and automated multicomponent SMS reminder system in improving referral uptake among schoolchildren in a low-resource setting.

Background:

Childhood visual impairment is common in low- and middle-income countries, but referral uptake after school-based vision screening remains poor. Mobile phone penetration and parents' use of messaging platforms provide an opportunity to use SMS-based interventions to improve follow-up care.

Objectives:

To assess the effectiveness of mHealth-based vision screening and SMS reminders on referral uptake among visually impaired children.

To explore the association of referral uptake with sociodemographic characteristics of children.

Methods:

This was a concurrent, parallel-group, single-blinded randomized controlled trial conducted in two Federal Government schools in Rawalpindi District, Pakistan. Children aged 5-15 years were screened for visual impairment using the validated Peek Acuity mobile application. Eligible children were randomized (school-level allocation, individual-level analysis) into two groups:

Intervention group: Received a printed referral form plus multicomponent SMS reminders (including health messages, visual depiction, practical action plan, and directions to hospital).

Control group: Received only the printed referral form (usual care).

Enrollment began on 21 October 2024 and was completed on 26 October 2024. Follow-up assessments continued for 8 weeks, with the last follow-up completed on 30 December 2024.

Sample size:

A total of 80 participants were enrolled, based on sample size calculations with adjustment for 10% expected dropout. Pilot testing on 8 additional participants (not included in the main analysis) ensured feasibility.

Blinding:

Due to the nature of the intervention, participants and field staff could not be blinded. However, outcome assessment (via weekly telephone follow-up) and data analysis were performed by independent researchers who were blinded to group assignment.

Outcomes:

Primary outcome: Proportion of referred children attending the hospital within 8 weeks.

Secondary outcome: Association of referral uptake with sociodemographic characteristics (e.g., age, sex, parental education).

Data collection and analysis:

Data were collected using the Peek-powered data collection platform, entered into encrypted devices, and analyzed with SPSS v27. An intention-to-treat approach was followed.

Ethics:

Ethical approval was obtained from the Ethical Review Committee, Army Medical College (NUMS). Permission to conduct the trial was provided by the FG Education Institutions Directorate, Rawalpindi. Written informed parental consent and child assent were required prior to participation.

Expected impact:

This trial is the first in Pakistan to evaluate the use of automated SMS reminders for improving referral uptake after school-based vision screening. Results will inform policymakers on how digital health interventions can strengthen child vision health services in resource-limited settings.

ELIGIBILITY:
Participants will only be enrolled if they meet all eligibility criteria:

* Age 5 to 15 years
* Detected with visual impairment on screening,
* Parent in possession of or have access to smartphone
* Parents have ability to receive, read and understand an SMS

Children may not enter the study if any of the following apply:

* Children with known refractive error (myopia)
* Children with spectacles
* Children with apparent eye diseases (e.g. conjunctivitis, red eye, ocular trauma, trachoma, etc.)
* Plan to travel outside the city in the next two months following enrollment

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Proportion of referred children who will attend the hospital within 8 weeks of referral in both groups | Follow up for 8 weeks on weekly basis after identification of visual impairment
  Primary outcome of interest is the proportion of referred children who attend the hospital within eight weeks of referral in both groups. It will be assessed by weekly telephonic follow up of referred children.

SECONDARY OUTCOMES:
Secondary outcome of interest is the association of hospital attendance with sociodemographic characteristics of referred participants | 1 - 56 day
  Secondary outcome of interest is the association of hospital attendance with sociodemographic characteristics of referred participants and will be assessed by comparing the sociodemographic characteristics of referred participants who attend the hospital with those who do not, using follow-up data.

CONTACTS AND LOCATIONS:
Overall Officials: Shamaila Mohsin, PhD, Study Director — National University of Medical Sciences
Locations (1):
- Federal government schools, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Javed A, Mohsin S. Effectiveness of mHealth-based vision screening on uptake of referral services among children of government schools in Rawalpindi, Pakistan: study protocol for a randomised controlled trial. BMJ Open. 2025 Oct 29;15(10):e096970. doi: 10.1136/bmjopen-2024-096970. PMID 41161831
- [Derived] Javed A, Mohsin S, Habib R, Malik UA. Effectiveness of mobile health based vision screening on uptake of referral services in school children: A randomized control trial. Pak J Med Sci. 2025 Aug;41(8):2328-2337. doi: 10.12669/pjms.41.8.11742. PMID 40980391
- See also: The Global Burden of Disease (GBD) study provides a comprehensive picture of mortality and disability across countries, time, age, and sex. — https://www.healthdata.org/research-analysis/gbd
- See also: Telecom Indicators, WHO fact sheet on blindness and visual impairment providing key facts, definitions, causes. — https://www.statista.com/statistics/262950/global-mobile-subscriptions-since-1993/
- See also: The IAPB Vision Atlas presents the very latest eye health data and evidence. — https://www.iapb.org/learn/vision-atlas/